CLINICAL TRIAL: NCT05570877
Title: A Multi-Centre, Randomized, 2-arm, Open-labelled, Controlled PMCF Study to Evaluate the Safety and Performance of ChitoCare Medical Wound Healing Gel in Healing of Chronic Wounds
Brief Title: ChitoCare Medical Wound Healing Gel PMCF Study on Healing of Chronic Wounds
Acronym: CHITOCHRONIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Primex ehf (Industry)
Collaborators: Vizera d.o.o. (Industry); University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHITOC-01
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer; Pressure Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Experimental): Active group will apply ChitoCare medical Wound Healing Gel to the wound in addition to standard of care.
  Interventions: Device: ChitoCare medical Wound Healing Gel
- Control group (No Intervention): Control group will only administer standard of care to treat their wounds.

INTERVENTIONS:
Device: ChitoCare medical Wound Healing Gel — ChitoCare medical Wound Healing Gel is a CE-marked medical device.
  Arms: Active group

SUMMARY:
We are testing a gel intended for the protection and healing of chronic wounds as a support for standard therapy. The main component of the gel is chitosan, a natural polymer that has the ability to stop bleeding, has a positive effect on wound healing, and has antimicrobial properties.

DETAILED DESCRIPTION:
The purpose of this PMCF study is to evaluate the safety and efficacy of ChitoCare medical Wound Healing Gel for the healing of chronic wounds. The study will enroll patients with diabetic foot ulcer, venous ulcer or pressure ulcer. Patients will be randomly assigned to an active or control group. The active group will apply the gel to the wound, in addition to the standard of care, while the control group will receive only standard care. The study will last from 3 to 18 months for an individual patient (15-month recruitment period and 3 months of follow-up after the last patient is enrolled) or until event occurrence (complete wound healing/exclusion from the study). The study envisages four visits: Visit 1 - Screening and Inclusion visit, Visit 2 (after 4 weeks), Visit 3 (after 12 weeks) and Visit 4 - End of Study Visit: The final visit will take place when the event occurs (complete healing/exclusion from study). On each visit, the patients will have their wound photographed and assessed after debridement. Adverse events will be followed throughout the whole study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be given
2. Patient ≥ 18 years old
3. Presence of chronic wound (Wagner grade I and II diabetic foot ulcer, venous leg ulcer or pressure ulcer) that meets the following criteria:

   * Size of the wound ≥ 0.5 cm2
   * Wound is not infected at the time of randomization
   * Wound is present for at least 4 weeks
4. Able to understand and comply with the requirements of the study

Exclusion Criteria:

1. Patients with serious concomitant disease (cancer, heart failure (NYHA class IV), severe anaemia (Hb<100 g/L), neoplasia)
2. Any significant condition that may preclude the participant from the study (e.g. severe depression or psychiatric illness)
3. Patients that will require surgical procedure to treat their ischemic condition on the limb where the wound is present as assessed by the investigator
4. Patients diagnosed with autoimmune connective tissue diseases
5. Previous treatment under this clinical protocol
6. Participation in another clinical trial
7. Receiving or scheduled to receive a medication or treatment which, in the opinion of the investigator, was known to interfere with, or affect the rate and quality of wound healing
8. Allergy to shellfish (for active study group)
9. Medical condition likely to require systemic corticosteroids during the study period
10. Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Time to complete healing | up to 18 months
  Hazard ratio for time to complete healing (active group vs. control group).

SECONDARY OUTCOMES:
Complete healing rate | 4 weeks, 12 weeks
  Proportion of completely healed ulcers (active group vs control group).
Reduction of wound size | 4 weeks, 12 weeks
  Relative reduction of wound surface area compared to baseline (active group vs control group).
Time to 75% and 50% healing | up to 18 months
  Hazard ratio for time to 75% and 50% healing
75% and 50% healing rate | 4 weeks, 12 weeks
  Proportion of 75% and 50% area healed ulcers (active group vs. control group)
Secondary infections | up to 18 months
  Occurrence of secondary infections
Incidence of adverse events (Safety of use) | up to 18 months
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Helene Liette Lauzon, Study Director — Primex ehf
Locations (9):
- Croatia (3):
  - Vuk Vrhovac University Clinic for Diabetes, Endocrinology and Metabolic Diseases, Merkur University Hospital, Zagreb, City of Zagreb
  - Clinical Hospital Sveti Duh, Zagreb
  - Marija Poliklinika, Zagreb
- Slovenia (6):
  - Medicina Mataln, Poljčane, Občina Poljčane
  - Ordinacija Andrej Kravos, Žalec, Občina Žalec
  - General Hospital Celje, Celje
  - Health Centre Koper, Koper
  - University Clinical Center Maribor, Maribor
  - Nursing Home Šmarje pri Jelšah, Šmarje pri Jelšah

IPD SHARING:
Plan to Share IPD: No